CLINICAL TRIAL: NCT00391040
Title: SGS: a Structured Treatment and Teaching Programme for Elderly Patients With Diabetes Mellitus - a Prospective Randomized Controlled Multicenter Trial
Brief Title: SGS: a Structured Treatment and Teaching Programme for Elderly Patients With Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Diabetes Association (Other)
Collaborators: Menarini Group (Industry); Deutsche Diabtesstiftung, Germany (Unknown)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 1201-10/03
Record Dates: First submitted 2006-10-20; First posted 2006-10-23 (Estimated); Last update posted 2006-10-23 (Estimated); Status verified 2006-10

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellitus, structured treatment and teaching, education,; elderly patients, geriatrics
MeSH Terms: conditions — Diabetes Mellitus

INTERVENTIONS:
Behavioral: SGS education

SUMMARY:
It was the aim of the study to develop and evaluate the effectiveness of a new structured teaching and training programme for elderly patients with diabetes mellitus (SGS) and insulin therapy.

DETAILED DESCRIPTION:
Patient education has become an integral part of any diabetes therapy in Germany. But elderly people are often not able to follow the variety of topics comprising standard treatment and training programmes for insulin-treated patients with type 2 diabetes mellitus due to geriatric syndromes and neuropsychological deficits. Therefore, treatment of elderly diabetics should focus on individual therapeutic goals, which reflect reduced life expectancy and quality of life.

It was the aim of the study to develop and evaluate the effectiveness of a new structured teaching and training programme for elderly patients with diabetes mellitus (SGS) and insulin therapy.

The high prevalence of cognitive impairment and affective disorders requires special pedagogical methods as well as adapted contents. For example the advantages of physical activity, the frequent existence of malnutrition, urinary incontinency or heart failure are taken into consideration. Contents are transmitted in a practical and daily-living oriented way.

The programme comprises 7 education lessons of 45 minutes duration implying the education units: diabetes mellitus, nutrition, treatment strategies, self-monitoring and complications focussing the diabetic foot syndrome.

The effectiveness of the new structured treatment and teaching programme SGS was evaluated in a multicenter prospective randomised controlled trial. Diabetic patients admitting one of 18 study centres in Germany with at least one geriatric syndrome, comorbidity and older than 65 years were randomised either to the new SGS programme or to the standard treatment programme for patients with type 2 diabetes mellitus. Before and 6 month after participation in the structured treatment programmes the outcome quality was evaluated using structured questionnaires. We assessed HbA1c, skills of diabetes self-management, diabetes knowledge, treatment satisfaction, acute and late complications, neuropsychological status, diabetes mediation, activities of daily living and need of social service. The main treatment goal was maintenance of autonomy and quality of life in elderly people, as well as prevention of catabolism, frailty and acute complications.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 65 years, at least more than one other diagnosis than diabetes, at least one geriatric syndrome

Exclusion Criteria:

* myocardial infarction, apoplexy within the last 2 weeks before planned enrolment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200
Dates: Start 2003-11; Study Completion 2006-05

PRIMARY OUTCOMES:
HbA1c decrease, reduction of hypoglycemia, acute complications

SECONDARY OUTCOMES:
treatment satisfaction, ability for diabetes management, diabetes knowledge

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Zeyfang, MD, Principal Investigator — German Diabetes Association- Working Group Diabetes and Geriatrics; Anke Braun, MD, Study Chair — German Diabetes Association- Working Group Diabetes and Geriatrics; Thomas Kubiak, MD, Study Chair — German Diabetes Association- Working Group Diabetes and Geriatrics; Ulrich A Müller, Prof, Study Chair — University of Jena; Jörn Kuntsche, MD, Study Chair — German Diabetes Association- Working Group Diabetes and Geriatrics; Martina Meier-Höfig, MD, Study Chair — German Diabetes Association- Working Group Diabetes and Geriatrics
Locations (1):
- Bethesda Hospital, Stuttgart, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Zeyfang A. [Diabetes in old age -- do we overstrain our patients?]. Dtsch Med Wochenschr. 2006 May 19;131(20):1159-62. doi: 10.1055/s-2006-941744. No abstract available. German. PMID 16705538
- [Result] Zeyfang A. [Structured educational programs for geriatric patients with diabetes mellitus]. MMW Fortschr Med. 2005 Jun 30;147(26):43, 45-6. German. PMID 16035489
- See also: a randomized controlled trial to proof effectiveness of a structured treatment and teaching programme for elderly patients with diabetes mellitus — http://www.diabetes-im-alter.de